CLINICAL TRIAL: NCT00000127
Title: Ischemic Optic Neuropathy Decompression Trial (IONDT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: NEI-26
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2009-09

CONDITIONS: Ischemic Optic Neuropathy
Keywords: Non-arteritic Ischemic Optic Neuropathy
MeSH Terms: conditions — Optic Neuropathy, Ischemic

INTERVENTIONS:
Procedure: Optic Nerve Sheath Decompression Surgery

SUMMARY:
To assess the safety and efficacy of optic nerve sheath decompression surgery for non-arteritic ischemic optic neuropathy (NAION).

DETAILED DESCRIPTION:
Non-arteritic ischemic optic neuropathy (NAION), the most common cause of acute optic nerve disease in older persons, causes permanent and severe visual loss. Visual function can be impaired through decreased central visual acuity or peripheral field loss, or both. NAION strikes both eyes in up to 40 percent of affected patients. The incidence of NAION has been estimated at 2.3 per 100,000 persons over the age of 50 years and 0.54 per 100,000 for all ages. Estimates of the number of new cases seen each year in the United States range from a low of approximately 1,500 to a high of 6,000.

NAION has been hypothesized to be caused by vascular insufficiency leading to optic nerve head ischemia. There is general agreement that NAION results from transient non-perfusion of nutrient vessels. The wide range of visual field defects and visual loss with NAION can be explained by the extent and number of the blood vessels involved.

Anatomical factors appear to contribute to the vascular event initiating NAION. Clinically, the number of discs congenitally lacking a physiological cup in eyes with NAION is higher than expected. Presumably, in eyes with NAION, these discs have small scleral openings that crowd the nerve fibers as they pass through the restricted space in the optic disc and lamina cribrosa, thereby predisposing to an ischemic spiral.

One current theory holds that NAION begins as a minor ischemic event that later progresses to a major infarction due to congenitally anomalous optic nerves. The inciting ischemic event leads to local anterior nerve edema, and this causes further ischemia.

Optic nerve sheath decompression surgery was reported in 1989 to be of benefit to patients with NAION. The presumed mechanism of action in optic nerve decompression surgery revolved around restoration of impaired blood flow to the optic nerve through reduction of the pressure around the nerve.

The Ischemic Optic Neuropathy Decompression Trial (IONDT) was a randomized clinical trial designed to compare the improvements in visual acuity at 6 months in patients assigned to receive surgery with optic nerve sheath decompression with those assigned to careful followup. A cohort of patients, with a baseline visual acuity of better than 20/64 are also being followed to better understand the natural history of the disease, including second eye involvement.

Enrollment began in October 1992. Randomization was stratified by clinic, and patients had an equal probability of assignment to surgery or careful followup. All patients are being followed for a minimum of 2 years.

The primary outcome is a change of three lines or more in visual acuity at the 6-month followup visit compared with visual acuity measured at the randomization visit.

Secondary outcomes include a change in visual acuity beyond 6 months, change in peripheral visual function as measured by automated Humphrey perimetry, local and systemic side effects from treatment, change in quality of life, and other associated morbidity and mortality.

ELIGIBILITY:
Men and women age 50 years or older, with acute NAION and visual symptoms for 14 days or less since the onset of symptoms, and visual acuity worse than or equal to 20/64 were eligible for randomization.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1992-10; Study Completion 1994-10 (Actual)

REFERENCES:
- [Background] The ischemic optic neuropathy decompression trial (IONDT): design and methods. Control Clin Trials. 1998 Jun;19(3):276-96. doi: 10.1016/s0197-2456(98)00003-8. PMID 9620811
- [Background] Characteristics of patients with nonarteritic anterior ischemic optic neuropathy eligible for the Ischemic Optic Neuropathy Decompression Trial. Arch Ophthalmol. 1996 Nov;114(11):1366-74. doi: 10.1001/archopht.1996.01100140566007. PMID 8906027
- [Background] Scherer RW; Crawley B; Abstracts for the Ischemic Optic Neuropathy Study Group; Responses to ethical and other questions on a knowledge assessment form for a multicenter trial. [Abstract]., Controlled Clinical Trials 1993;14:442S
- [Background] Crawley B; Scherer RW; Ischemic Optic Neuropathy Decompression Trial (IONDT): Participation in the IONDT. Race, gender and age. [Abstract]., Controlled Clinical Trials 1994;15:102S
- [Background] Crawley B; Waring MT; Scherer RW; Coordinating Center for the Ischemic Optic Neuropathy Decompression Trial (IONDT): IONDT tracking system: Where is form 2034 for patient ICMORE and who is responsible? [Abstract]., Controlled Clinical Trials 1994;15:93S
- [Background] Optic nerve decompression surgery for nonarteritic anterior ischemic optic neuropathy (NAION) is not effective and may be harmful. The Ischemic Optic Neuropathy Decompression Trial Research Group. JAMA. 1995 Feb 22;273(8):625-32. PMID 7844872